CLINICAL TRIAL: NCT03470961
Title: Safety and Efficacy of Polyclonal Antibodies in Simultaneous Pancreas Kidney Transplant Recipients: Single-centre, Prospective, Observational Study
Brief Title: Observational Study to Evaluate the Safety and Efficacy of Polyclonal Antibodies in Simultaneous Pancreas Kidney Transplant Recipients
Acronym: PAISPK
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin First Central Hospital (Other)
Responsible Party: Principal Investigator, Yingxin FU.MD, Head of Department, Tianjin First Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018N017KY
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: CKD (Chronic Kidney Disease) Stage 5T; Diabetes Mellitus; Simultaneous Pancreas Kidney Transplantation
Keywords: Grafalon ATG SPK
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus | interventions — Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-Tlymphocyte Globulins (Experimental): intravenous，2mg/kg/d，for 5 days
  Interventions: Drug: Anti-Tlymphocyte Globulins
- Anti-thymocyte Globulins (Active Comparator): intravenous，1.5mg/kg/d，for 4 days
  Interventions: Drug: Anti-Thymocyte Globulins

INTERVENTIONS:
Drug: Anti-Tlymphocyte Globulins — Induction therapy regimen in simultaneous pancreas kidney transplantation
  Other Names: Grafalon; ATG-F
  Arms: Anti-Tlymphocyte Globulins
Drug: Anti-Thymocyte Globulins — Induction therapy regimen in simultaneous pancreas kidney transplantation
  Other Names: ATG
  Arms: Anti-thymocyte Globulins

SUMMARY:
A single-centre, prospective, observational study to evaluate the safety and efficacy of Polyclonal Antibodies in simultaneous Pancreas Kidney Transplant recipients.

DETAILED DESCRIPTION:
Polyclonal antibody mainly contains Antit-Tlymphocyte globulins(Grafalon) and Anti-thymocyte globulins(ATG). To investigate the efficacy and safety of polyclonal antibodies induction regimen using Grafalon compared with ATG in de novo simultaneous pancreas kidney transplant recipients. The primary analysis of this study is to demonstrate the non-inferiority of the two regimens with regard to efficacy, defined as failure rate.

The secondary objective of the study is the assessment of safety and further efficacy parameters in terms of incidence of acute rejections, graft/patient survival, DGF(delayed graft function), pancreas function and renal function

ELIGIBILITY:
Inclusion Criteria:

1. with end-stage,diabetic nephropathy(type1or 2)
2. Patients scheduled to undergo SPK with compatible ABO blood type.
3. Peak PRA <50%
4. Females of childbearing potential must have a negative pregnancy test within 48hrs prior to randomization and reliable methods of contraception should be started 4 weeks prior to and during the whole study.
5. Patient must have signed the Patient Informed Consent Form.
6. Patient must receive a primary simultaneous pancreas/kidney (SPK) cadaveric transplant, with either intestinal or bladder and either portal or systemic venous drainages.

Exclusion Criteria:

1. Patient is pregnant or breastfeeding.
2. Patient has a positive T-cell crossmatch on the most recent serum specimen.
3. Patient is known for active liver disease or has significant liver disease, defined by ASAT and ALAT serum levels greater than 3 times the upper limit of normal.
4. Patient has malignancy or history of malignancy, with the exception of adequately treated localised squamous cell or basal cell carcinoma, without recurrence.
5. Patient has been included in another clinical trial protocol for any investigational drug within 4 weeks prior to randomisation.
6. Patient has any form of substance abuse, psychiatric disorder or condition, which, in the opinion of the investigator, may invalidate communication.
7. Patient receives a SPK transplant from a living donor, or receives segmental pancreatic transplant, or a previous kidney transplant alone.
8. Donor is older than 55 years of age
9. patients with bacterial, viral or mycotic infections which are not under therapeutically control

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse event | up to 3 months post-transplantation
  Incidence of patient's death,graft loss,acute rejection

CONTACTS AND LOCATIONS:
Overall Officials: Yingxin FU, M.D, Principal Investigator — Tianjin First Central Hospital
Locations (1):
- Tianjin First central hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Burkhalter F, Schaub S, Bucher C, Gurke L, Bachmann A, Hopfer H, Dickenmann M, Steiger J, Binet I. A Comparison of Two Types of Rabbit Antithymocyte Globulin Induction Therapy in Immunological High-Risk Kidney Recipients: A Prospective Randomized Control Study. PLoS One. 2016 Nov 17;11(11):e0165233. doi: 10.1371/journal.pone.0165233. eCollection 2016. PMID 27855166
- [Result] Kuypers DR, Malaise J, Claes K, Evenepoel P, Maes B, Coosemans W, Pirenne J, Vanrenterghem Y; Euro-SPK Study Group. Secondary effects of immunosuppressive drugs after simultaneous pancreas-kidney transplantation. Nephrol Dial Transplant. 2005 May;20 Suppl 2:ii33-9, ii62. doi: 10.1093/ndt/gfh1080. PMID 15814548